CLINICAL TRIAL: NCT05402995
Title: Prospective Randomized Control Trial Comparing Irrisept to Saline Irrigation for the Prevention of Infection After Open Tibia Fractures
Brief Title: Randomized Trial Comparing Irrisept to Saline Irrigation for Infection Prevention
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was not progressing as expected.
Sponsor: Brett D. Crist (Other)
Responsible Party: Sponsor-Investigator, Brett D. Crist, Professor, Director Orthopaedic Trauma Service, Director Orthopaedic Trauma Fellowship, Surgery of the Hip and Trauma, Department of Orthopaedic Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2086908
Record Dates: First submitted 2022-04-05; First posted 2022-06-02 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Gustilo-Anderson Type III Open Tibia Fracture
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled and randomized into one of four groups:
  1. Standard operative debridement and spanning external fixator (reference/control group)
  2. Spanning external fixator with Irrisept irrigation (treatment group 1)
  3. Antibiotic-coated medullary nail with saline irrigation (treatment group 2) or
  4. Antibiotic-coated medullary nail with Irrisept irrigation (treatment group 3)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard operative debridement and spanning external fixator (reference/control group) (Active Comparator): This is the standard of care management. Patient will go to the operating room (OR) first for irrigation and debridement with normal saline and external fixation. Will return to OR at a later date for definitive fixation.
  Interventions: Drug: Saline
- Spanning external fixator with Irrisept irrigation (treatment group 1) (Experimental): Patient will go to the operating room (OR) first for irrigation and debridement with Irrisept (the experimental irrigation solution) and external fixation. Will return to OR at a later date for definitive fixation.
  Interventions: Drug: Irrisept (Irrigation Solution)
- Antibiotic-coated medullary nail with saline irrigation (treatment group 2) (Experimental): Patient will go to the operating room (OR) for treatment with an antibiotic-coated nail and have irrigation and debridement with normal saline.
  Interventions: Drug: Saline
- Antibiotic-coated medullary nail with Irrisept irrigation (treatment group 3) (Experimental): Patient will go to the operating room (OR) for treatment with an antibiotic-coated nail and have irrigation and debridement with Irrisept (the experimental irrigation solution).
  Interventions: Drug: Irrisept (Irrigation Solution)

INTERVENTIONS:
Drug: Irrisept (Irrigation Solution) — Irrisept Antimicrobial Wound Lavage is intended for mechanical cleansing and removal of debris, dirt and foreign materials, including microorganisms from wounds.
  Arms: Antibiotic-coated medullary nail with Irrisept irrigation (treatment group 3); Spanning external fixator with Irrisept irrigation (treatment group 1)
Drug: Saline — Saline irrigation
  Arms: Antibiotic-coated medullary nail with saline irrigation (treatment group 2); Standard operative debridement and spanning external fixator (reference/control group)

SUMMARY:
Early debridement and definitive fixation, at the initial operative setting, historically led to no difference in the infection rates for Gustilo-Anderson type III open tibia fractures. However, Lenarz et al. reported that delaying definitive fixation in open tibia fractures could decrease the deep infection rate. At the University of Missouri, the investigators found that staged procedures, including initial debridement-temporary fixation and delayed definitive fixation, did not statistically decrease the rate of deep infection in Gustilo-Anderson type III fractures, prompting the study that is being proposed here. Antibiotic cement coated intramedullary nails have been used in management of infected long bone fractures. Since external fixation and staged debridement did not decrease type III open tibia infection rate, the investigators wanted to consider using antibiotic cement coated nails to deliver antibiotics locally in the acute open fracture setting to prophylactically decrease associated infection rate. Additionally, Irrisept is a wound irrigant that has been used to lower infection rates in different wound settings. To the investigators' knowledge, there are no robust data showing its effectiveness at lowering infection rates in open tibia fracture management. The purpose of this study is to determine the effects of Irrisept and antibiotic nails on lowering deep infection rates in type III open tibia fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, 18 or over
2. Gustilo-Anderson type III open tibia fracture
3. Able to obtain informed consent from patient

Exclusion Criteria:

1. Minor, under 18
2. Pregnancy
3. Prisoner
4. Allergic to chlorhexidine gluconate
5. Allergic to vancomycin or tobramycin
6. Patient's tibia is unable to accommodate the smallest antibiotic nail
7. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Operative Debridement and Spanning External Fixator (Reference/Control Group) | Spanning External Fixator With Irrisept Irrigation (Treatment Group 1) | Antibiotic-coated Medullary Nail With Saline Irrigation (Treatment Group 2) | Antibiotic-coated Medullary Nail With Irrisept Irrigation (Treatment Group 3)
Started | 0 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 2 | 2
Not completed — Study terminated due to lack of enrollment and followup. | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: As study was terminated due to difficulty enrolling participants there was no one randomized to the reference/control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Operative Debridement and Spanning External Fixator (Reference/Control Group) | Spanning External Fixator With Irrisept Irrigation (Treatment Group 1) | Antibiotic-coated Medullary Nail With Saline Irrigation (Treatment Group 2) | Antibiotic-coated Medullary Nail With Irrisept Irrigation (Treatment Group 3) | Total
Number analyzed (Participants) | 0 | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2 | 1 | 5
  >=65 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1
  Male | 0 | 2 | 2 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Surgical Site Infection (SSI)
Description: Measured by the number of surgical site infections in the total population of patients.
Time Frame: 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Operative Debridement and Spanning External Fixator (Reference/Control Group) | Spanning External Fixator With Irrisept Irrigation (Treatment Group 1) | Antibiotic-coated Medullary Nail With Saline Irrigation (Treatment Group 2) | Antibiotic-coated Medullary Nail With Irrisept Irrigation (Treatment Group 3)
Number analyzed (Participants) | 0 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Fracture Healing
Description: Presence or absence of fracture callous measured on x-ray by an experienced orthopaedic surgeon.
Time Frame: 6 months
Population: As study was terminated due to difficulty enrolling participants there was no one randomized to the reference/control group. Unable to measure presence or absence of fracture callus due to lack of follow-up with study termination.
Arm/Group | Standard Operative Debridement and Spanning External Fixator (Reference/Control Group) | Spanning External Fixator With Irrisept Irrigation (Treatment Group 1) | Antibiotic-coated Medullary Nail With Saline Irrigation (Treatment Group 2) | Antibiotic-coated Medullary Nail With Irrisept Irrigation (Treatment Group 3)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: There is a minimal increased risk of reaction to chlorhexidine gluconate in the Irrisept treatment group which may include allergic reaction or irritation therefore adverse event / serious adverse events are not anticipated and would be considered a result of the injury sustained.
Arm/Group | Standard Operative Debridement and Spanning External Fixator (Reference/Control Group) | Spanning External Fixator With Irrisept Irrigation (Treatment Group 1) | Antibiotic-coated Medullary Nail With Saline Irrigation (Treatment Group 2) | Antibiotic-coated Medullary Nail With Irrisept Irrigation (Treatment Group 3)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Operative Debridement and Spanning External Fixator (Reference/Control Group) (N=0) | Spanning External Fixator With Irrisept Irrigation (Treatment Group 1) (N=2) | Antibiotic-coated Medullary Nail With Saline Irrigation (Treatment Group 2) (N=2) | Antibiotic-coated Medullary Nail With Irrisept Irrigation (Treatment Group 3) (N=2)
Amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT05402995/Prot_SAP_000.pdf